CLINICAL TRIAL: NCT05292391
Title: A Phase 1, Open-Label, Dose-Escalation Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Sm-p80 + GLA-SE (SchistoShield(R)) Vaccine in Healthy Adults
Brief Title: Safety, Tolerability, and Immunogenicity Study of Sm-p80 + GLA-SE (SchistoShield(R)) Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 18-0018; 5UM1AI148373-03 (NIH)
Record Dates: First submitted 2022-03-03; First posted 2022-03-23 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-10-30

CONDITIONS: Schistosomiasis
Keywords: Dose-Escalation; Immunigenicity; Open-label; Phase I; Reactogenicity; Schistosomiasis; Vaccine
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- A (Experimental): 0.5 mL of 100 micrograms of Sm-p80 administered intramuscularly on Days 1, 29, and 57. N=9
  Interventions: Biological: Sm-p80
- B (Experimental): 0.5 mL of 10 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57. N=9
  Interventions: Biological: Sm-p80 + GLA-SE
- C (Experimental): 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 180. N=9.
  Interventions: Biological: Sm-p80 + GLA-SE
- D (Experimental): 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57. N=9.
  Interventions: Biological: Sm-p80 + GLA-SE
- E (Experimental): 0.5mL of 100 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29 and 57. N=9.
  Interventions: Biological: Sm-p80 + GLA-SE

INTERVENTIONS:
Biological: Sm-p80 — The Sm-p80 protein is formulated and lyophilized to yield the vaccine antigen, Sm-p80 for Injection.
  Arms: A
Biological: Sm-p80 + GLA-SE — Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.
  Arms: B; C; D; E

SUMMARY:
This is a Phase 1, open-label, dose-escalation clinical trial to evaluate the safety, reactogenicity, and immunogenicity of the Sm-p80+GLA-SE vaccine candidate in healthy adults between 18 and 55 years of age. Forty-five subjects will receive a series of three intramuscular injections 28 days apart with dose based on group. Five treatment groups, each including nine subjects, will receive three intramuscular (IM) injections of 0.5 mL of the designated study product on either Days 1, 29, and 57 or on Days 1, 29, and 180 (Table 1). Group A (unadjuvanted comparator) will receive 100 micrograms Sm-p80 alone on Days 1, 29, and 57, Group B (low dose standard schedule) will receive 10 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 57, Group C (mid dose delayed booster) will receive 30 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 180, Group D (mid dose standard schedule) will receive 30 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29, and 57, and Group E (high dose standard schedule) will receive 100 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 57. Study duration is approximately 20 months and will be conducted at one site in the US. Participant duration for subjects is 15 months. The primary objective is to assess the safety and reactogenicity following receipt of three doses of 1) 100 micrograms Sm- p80 (unadjuvanted), 2) 10 micrograms Sm-p80 + 5 micrograms GLA-SE, 3) 30 micrograms Sm-p80 + 5 micrograms GLA- SE, and 4) 100 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57 and 5) 30 micrograms Sm-p80 + 5 micrograms GLA- SE administered on Days 1, 29, and 180.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalation clinical trial to evaluate the safety, reactogenicity, and immunogenicity of the Sm-p80+GLA-SE vaccine candidate in healthy adults between 18 and 55 years of age. Forty-five subjects will receive a series of three intramuscular injections 28 days apart with dose based on group. Five treatment groups, each including nine subjects, will receive three intramuscular (IM) injections of 0.5 mL of the designated study product on either Days 1, 29, and 57 or on Days 1, 29, and 180 (Table 1). Group A (unadjuvanted comparator) will receive 100 micrograms Sm-p80 alone on Days 1, 29, and 57, Group B (low dose standard schedule) will receive 10 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 57, Group C (mid dose delayed booster) will receive 30 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 180, Group D (mid dose standard schedule) will receive 30 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29, and 57, and Group E (high dose standard schedule) will receive 100 micrograms Sm-p80 + 5 micrograms GLA-SE on Days 1, 29 and 57. Study duration is approximately 20 months and will be conducted at one site in the US. Participant duration for subjects is 15 months. The primary objective is to assess the safety and reactogenicity following receipt of three doses of 1) 100 micrograms Sm- p80 (unadjuvanted), 2) 10 micrograms Sm-p80 + 5 micrograms GLA-SE, 3) 30 micrograms Sm-p80 + 5 micrograms GLA- SE, and 4) 100 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57 and 5) 30 micrograms Sm-p80 + 5 micrograms GLA- SE administered on Days 1, 29, and 180. The secondary objectives are to assess anti- Sm-p80 Immunoglobulin G (IgG) antibody responses for all subjects from samples collected at specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 18 through 55 years of age, inclusive, at the time of consent.
2. Able and willing to participate for the duration of the study and able to understand and comply with planned study procedures.
3. Able and willing to provide written (not proxy) informed consent.
4. Is in good health, as judged by the investigator, and determined by medical history and physical examination*.

   *Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable. A stable medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last three months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last six months (180 days). Any change due to change of health care provider, insurance company, or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site PI or appropriate sub-investigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of solicited events and immunogenicity. Topical, nasal, and inhaled medications (with the exception of some uses of corticosteroids as outlined in the Subject Exclusion Criteria), vitamins, and contraceptives are permitted.
5. Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study product injection.

   *Not sterilized via bilateral tubal ligation, bilateral oophorectomy, or hysterectomy, or, if menopausal, still menstruating or < 1 year of the last menses
6. Women of childbearing potential must have used an acceptable form of contraception* in the 30 days prior to their first study product injection.

   *Acceptable single forms of contraception include abstinence from sexual activity that could lead to pregnancy, monogamous relationship with vasectomized partner who has been vasectomized for six months or more prior to enrollment, successful Essure placement (permanent, non-surgical, non-hormonal sterilization), intrauterine devices, and hormonal methods, including the birth control patch, shot (Depo-Provera), pills, the vaginal ring (NuvaRing), and the contraceptive implant (Nexplanon). Acceptable barrier methods include diaphragm or cervical cap with spermicide and the contraceptive sponge.
7. Women of childbearing potential must agree to continue use of an acceptable form of contraception through 30 days after their last study product injection.
8. Weight >/= 50 kg and body mass index (BMI) < 35.0 kg/m2
9. Vital signs (oral temperature, pulse, and blood pressure) are all within normal protocol-defined ranges.*

   *The normal protocol-defined ranges for vital signs include (a) oral temperature less than 38 degrees C (100.4 degrees F), (b) pulse no greater than 100 bpm, (c) systolic blood pressure 85 to 150 mmHg, inclusive, and (d) diastolic BP </= 100 mmHg.
10. Screening clinical lab values are all within normal protocol-defined reference ranges.

    * The normal protocol-defined ranges for laboratory tests include (a) ALT of < 47 IU/L, (b) creatinine less than or equal to the laboratory upper limit of normal, (c) WBC >/=3.80 x10^3/UL and </=13.00 x10^3/UL, (d) hemoglobin 11.5 g/dL or greater for females or 12.6 g/dL or greater for males, (e) platelets between 131 x10^3/UL and 415 x10^3/UL, inclusive.

Exclusion Criteria:

1. Has had known schistosomiasis infection or has traveled to an endemic area for schistosomiasis infection and, during that travel, was potentially exposed to a Schistosoma species.
2. Has been treated for schistosomiasis.
3. Has previous exposure to schistosome vaccines or experimental products containing GLA-SE.
4. Female subjects who are breastfeeding a child ,or who plan to breastfeed a child from the first study product injection through 30 days after the last study product injection.
5. Asthma, other than mild, well-controlled asthma*

   *Cold or exercise-induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Subjects should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year
6. Known atherosclerotic cardiovascular disease or history of myocardial infarction, pericarditis, or myocarditis.
7. Diabetes mellitus
8. History of a psychiatric condition that may make study compliance difficult, such as schizophrenia, or poorly controlled bipolar disorder**

   **Includes persons with psychoses or history of suicide attempt or gesture in the 3 years before study entry or an ongoing risk for suicide.
9. Chronic or active neurologic condition (including seizures*** and migraine headaches****).

   ***Seizure within the past 5 years

   ****Four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care.
10. Autoimmune disease******

    ******autoimmune hypothyroidism with or without replacement therapy, and vitiligo or mild eczema or psoriasis not requiring chronic therapy, are permissible
11. Known or suspected congenital or acquired immunodeficiency including anatomic or functional asplenia******* or immunosuppression as a result of underlying illness or treatment.

    *******Any splenectomy is exclusionary.
12. Use of alcohol or drugs that, in the opinion of the investigator, may interfere with ability to comply with the protocol or increase risk to subject's health during the study period.
13. Active neoplastic disease********

    ********Subjects with a history of malignancy may be included if treated by surgical excision, or by chemotherapy or radiation therapy and has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months). Cervical neoplasia under surveillance and non-melanoma skin cancer are not exclusionary.
14. Chronic topical or systemic corticosteroid use*********

    *********Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis prior to enrollment may be enrolled the day after their therapy is completed. Oral or parenteral (intravenous, IM, subcutaneous) corticosteroids given for non-chronic conditions not expected to recur are permissible if, within the year prior to enrollment, the longest course of therapy was no more than 14 days and no oral or parenteral corticosteroids were given within 30 days prior to enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was at least 30 days prior to enrollment. Topical or systemic corticosteroid use for study related AEs is not exclusionary.
15. Known contraindication to repeated phlebotomy**********

    **********Such as minimal venous access or recent history of anemia
16. Receipt or planned receipt of inactivated vaccine or allergy desensitization injection within 14 days before or after a study product injection.
17. Receipt or planned receipt of live attenuated vaccine within 28 days before or after a study product injection.
18. Receipt of blood products or immunoglobulin within six months prior to, or donation of a unit of blood within two months prior to, the first study product injection.
19. Receipt of any experimental agent*********** within 30 days prior to screening or planned receipt prior to the last study visit-**.

    ***********Vaccine, drug, biologic, device, blood product, or medication.

    **Receipt of experimental COVID-19 related products are not necessarily exclusionary and will be evaluated on a case-by-case basis.
20. Plan to undergo surgery (elective or otherwise) within six months after study enrollment.
21. Plans to enroll in another interventional clinical trial************ at any time during the study period.

    ************Includes trials evaluating interventions such as a drug, biologic, or device.
22. Positive confirmatory test for HIV infection.
23. Positive serologic test for hepatitis B surface antigen (HBsAg).
24. Positive confirmatory test for hepatitis C virus (HCV) infection.
25. Acute febrile illness (oral temperature = 38°C) or other acute illness within three days prior to study product injection.*************

    *************Note for afebrile, acute illness only: If a subject is afebrile, his/her acute illness is nearly resolved with only minor residual symptoms remaining, and, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol, the subject may receive study product injection without further approval from the DMID Medical Officer.
26. Not willing to avoid donating blood during the study.
27. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Jackson LA, Coler RN, Deye GA, Carter D, Gray SA, Pecor T, Davis J, Larsen SE, Posavad CM, Cox C, Watanabe A, Lundeen JS, Gill R, Kalyanasundaram A, Siddiqui AA. Safety and immunogenicity of the Sm-p80 GLA-SE schistosomiasis vaccine. NPJ Vaccines. 2025 Nov 24;10(1):247. doi: 10.1038/s41541-025-01261-3. PMID 41285840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population includes 45 healthy adults ages 18 through 55 years who met all eligibility criteria. Participants were enrolled between 23May2022 to 24Jan2023.
Groups:
- Group A: 100 ug Sm-p80 Unadjuvanted: 0.5 mL of 100 micrograms of Sm-p80 administered intramuscularly on Days 1, 29, and 57.
  Sm-p80: The Sm-p80 protein is formulated and lyophilized to yield the vaccine antigen, Sm-p80 for Injection.
- Group B: 10 ug Sm-p80 + GLA-SE: 0.5 mL of 10 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57.
  Sm-p80 + GLA-SE: Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.
- Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster: 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 180.
  Sm-p80 + GLA-SE: Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.
- Group D: 30 ug Sm-p80 + GLA-SE: 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57.
  Sm-p80 + GLA-SE: Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.
- Group E: 100 ug Sm-p80 + GLA-SE: 0.5mL of 100 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29 and 57.
  Sm-p80 + GLA-SE: Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.
Period: Overall Study
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Started | 9 | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: 100 ug Sm-p80 Unadjuvanted: 0.5 mL of 100 micrograms of Sm-p80 administered intramuscularly on Days 1, 29, and 57.
- Group B: 10 ug Sm-p80 + GLA-SE: 0.5 mL of 10 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57.
- Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster: 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 180.
- Group D: 30 ug Sm-p80 + GLA-SE: 0.5mL of 30 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29, and 57.
- Group E: 100 ug Sm-p80 + GLA-SE: 0.5mL of 100 micrograms Sm-p80 + 5 micrograms GLA-SE administered intramuscularly on Days 1, 29 and 57.
- Total: Total of all reporting groups
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.2) | 40.8 (10.0) | 35.4 (7.3) | 34.0 (9.9) | 38.8 (13.0) | 37.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7 | 6 | 6 | 26
  Male | 6 | 5 | 2 | 3 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 9 | 9 | 7 | 8 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 8 | 8 | 8 | 6 | 8 | 38
  More than one race | 1 | 0 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 9 | 45
Height [Mean (Standard Deviation); unit: cm] | 169.58 (6.23) | 175.19 (7.50) | 168.14 (9.28) | 166.62 (5.67) | 171.33 (6.63) | 170.17 (7.46)
Weight [Mean (Standard Deviation); unit: kg] | 75.62 (13.94) | 77.89 (10.35) | 72.81 (11.38) | 73.59 (12.40) | 71.68 (13.27) | 74.32 (11.97)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.27 (4.34) | 25.29 (2.00) | 25.72 (3.38) | 26.46 (3.99) | 24.39 (4.06) | 25.62 (3.56)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Throughout the Study
Description: An AE or suspected adverse reaction were considered an SAE if, in the view of either the principal investigator or the sponsor, resulted in any of the following outcomes:
  * Death,
  * A life-threatening AE,
  * Inpatient hospitalization or prolongation of existing hospitalization,
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
  * A congenital anomaly/birth defect.
  * Important medical events that may not have resulted in death, been life-threatening, or required hospitalizations could have been considered serious when, based upon appropriate medical judgment they could have jeopardized the patient or participant and may have required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Through 12 months after the last study vaccination. For Groups A, B, D, E: Day 1 through Day 422. For Group C: Day 1 through Day 545
Population: The safety population includes all participants who received at least one dose of the study product and is summarized according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Solicited Reactogenicity Events Within 7 Days Post Each Dose
Description: Systemic symptoms collected include arthralgia, chills, fatigue, fever, headache, malaise, myalgia, nausea, and vomiting.
  Injection site (local) symptoms collected include erythema/redness (measurement), induration/swelling (functional and measurement), pain, pruritus, and tenderness
Time Frame: For Groups A, B, D, E: Post Dose 1 Day 1 through Day 8, Post Dose 2 Day 29 through Day 36, Post Dose 3 Day 57 through 64. For Group C: Post Dose 1 Day 1 through Day 8, Post Dose 2 Day 29 through 36, Post Dose 3 Day 180 through Day 187.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants
  Post Dose 1 | 9 | 9 | 8 | 5 | 9
  Post Dose 2: number analyzed (Participants) | 9 | 9 | 9 | 7 | 8
  Post Dose 2 | 9 | 7 | 8 | 7 | 6
  Post Dose 3: number analyzed (Participants) | 9 | 9 | 9 | 7 | 8
  Post Dose 3 | 8 | 9 | 9 | 7 | 7

3. Primary Outcome: Number of Participants Reporting Chemistry Laboratory Adverse Events (AEs) Within 28 Days Post Each Dose
Description: Chemistry measurements collected include alanine aminotransferase (ALT) and creatinine.
  Labs were collected on vaccination days and 7 days and 28 days post each vaccination.
Time Frame: Through 28 days after each study vaccination. For Groups A, B, D, E: Day 1 through Day 85. For Group C: Day 1 through Day 57, Day 180 through Day 208
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants
  Day 1: No events | 9 | 9 | 8 | 9 | 9
  Day 1: Mild events | 0 | 0 | 1 | 0 | 0
  Day 8: No events | 9 | 9 | 9 | 9 | 9
  Day 8: Mild events | 0 | 0 | 0 | 0 | 0
  Day 29: number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
  Day 29: No events | 9 | 9 | 9 | 8 | 9
  Day 29: Mild events | 0 | 0 | 0 | 0 | 0
  Day 36: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  Day 36: No events | 8 | 9 | 9 | 8 | 8
  Day 36: Mild events | 1 | 0 | 0 | 0 | 0
  Day 57: number analyzed (Participants) | 9 | 9 | 9 | 9 | 8
  Day 57: No events | 9 | 9 | 9 | 9 | 8
  Day 57: Mild events | 0 | 0 | 0 | 0 | 0
  Day 64: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 64: No events | 9 | 9 |  | 8 | 8
  Day 64: Mild events | 0 | 0 |  | 0 | 0
  Day 85: number analyzed (Participants) | 8 | 9 | 0 | 8 | 8
  Day 85: No events | 8 | 9 | 0 | 7 | 8
  Day 85: Mild events | 0 | 0 | 0 | 1 | 0
  Day 180: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 180: No events |  |  | 9 |  |
  Day 180: Mild events |  |  | 0 |  |
  Day 187: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 187: No events |  |  | 9 |  |
  Day 187: Mild events |  |  | 0 |  |
  Day 208: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 208: No events |  |  | 9 |  |
  Day 208: Mild events |  |  | 0 |  |

4. Primary Outcome: Number of Participants Reporting Hematology Laboratory Adverse Events (AEs) Within 28 Days Post Each Dose
Description: Hematology measurements include white blood cells (WBC), hemoglobin, and platelets.
  Labs were collected on vaccination days and 7 days and 28 days post each vaccination.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants
  Day 1: No events | 9 | 9 | 9 | 9 | 9
  Day 1: Mild or Moderate Events | 0 | 0 | 0 | 0 | 0
  Day 8: number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
  Day 8: No events | 8 | 6 | 9 | 9 | 8
  Day 8: Mild or Moderate Events | 0 | 3 | 0 | 0 | 1
  Day 29: number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
  Day 29: No events | 8 | 9 | 9 | 8 | 8
  Day 29: Mild or Moderate Events | 1 | 0 | 0 | 0 | 1
  Day 36: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  Day 36: No events | 9 | 8 | 9 | 8 | 7
  Day 36: Mild or Moderate Events | 0 | 1 | 0 | 0 | 1
  Day 57: number analyzed (Participants) | 9 | 9 | 9 | 9 | 8
  Day 57: No events | 9 | 9 | 7 | 9 | 7
  Day 57: Mild or Moderate Events | 0 | 0 | 2 | 0 | 1
  Day 64: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 64: No events | 9 | 8 |  | 8 | 6
  Day 64: Mild or Moderate Events | 0 | 1 |  | 0 | 2
  Day 85: number analyzed (Participants) | 8 | 9 | 0 | 8 | 8
  Day 85: No events | 8 | 7 |  | 7 | 8
  Day 85: Mild or Moderate Events | 0 | 2 |  | 1 | 0
  Day 180: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 180: No events |  |  | 9 |  |
  Day 180: Mild or Moderate Events |  |  | 0 |  |
  Day 187: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 187: No events |  |  | 9 |  |
  Day 187: Mild or Moderate Events |  |  | 0 |  |
  Day 208: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 208: No events |  |  | 8 |  |
  Day 208: Mild or Moderate Events |  |  | 1 |  |

5. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs) Within 28 Days Post Each Dose
Description: Unsolicited adverse events (AEs) were defined as an untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Unsolicited AEs do not include solicited events that began within the reactogenicity period (7 days post dose).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
participants
  Related Mild Events | 1 | 2 | 0 | 1 | 3
  Related Moderate Events | 1 | 1 | 0 | 1 | 0
  Related Severe Events | 0 | 0 | 0 | 0 | 0
  Not Related Mild Events | 3 | 6 | 2 | 6 | 2
  Not Related Moderate Events | 6 | 1 | 7 | 0 | 3
  Not Related Severe Events | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), New Onset Chronic Medical Condition (NOCMCs), and Potentially Immune-mediated Medical Conditions (PIMMCs)
Description: SAEs were AEs that resulted in any of the following: Death, Life-threatening, Hospitalization, Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, Congenital anomaly/birth defect. Important medical events based upon appropriate medical judgment they could have jeopardized the participant and may have required intervention to prevent one of the outcomes listed. MAAEs were hospitalization, ER visit, or an otherwise unscheduled visit to or from medical personnel for any reason and considered related to study product. NOCMCs were any new ICD-10 diagnosis that applied to the participant during the duration of the study, after receipt of the study agent, that was expected to continue for at least 3 months and require continued health care intervention. PIMMCs were AEs that include diseases which are clearly autoimmune in etiology and other inflammatory and/or neurologic disorders which may or may not have autoimmune etiologies.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants
  SAE | 0 | 0 | 0 | 0 | 0
  MAAE | 0 | 0 | 0 | 0 | 0
  NOCMC | 1 | 0 | 0 | 0 | 0
  PIMMC | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Achieving Seroconversion in Sm-p80 IgG Antibodies 28 Days Post Each Dose
Description: Seroconversion was defined as a fourfold rise from baseline.
Time Frame: Through 28 days after the first, second, and third study vaccinations. For Groups A, B, D, E: Day 8, 29, 36, 57, 64, and Day 85. For Group C: Day 8, 29, 36, 57, 180, 187, and Day 208.
Population: The modified intention-to-treat (mITT) immunogenicity population includes all participants who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination venous blood sample for immunogenicity testing for which valid results were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Participants
  Day 8 | 0 | 0 | 0 | 0 | 0
  Day 29: number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
  Day 29 | 1 | 0 | 2 | 1 | 2
  Day 36: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  Day 36 | 4 | 6 | 8 | 7 | 8
  Day 57: number analyzed (Participants) | 9 | 9 | 9 | 9 | 8
  Day 57 | 5 | 8 | 8 | 7 | 8
  Day 64: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 64 | 8 | 9 |  | 7 | 8
  Day 85: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 85 | 8 | 9 |  | 7 | 8
  Day 180: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 180 |  |  | 6 |  |
  Day 187: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 187 |  |  | 8 |  |
  Day 208: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 208 |  |  | 8 |  |

8. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Sm-p80 IgG Antibodies 7 Days and 28 Days Post Each Dose and 124 Days Post Dose 3
Description: Geometric mean titers (GMTs).
Time Frame: Through 7 and 28 days after each vaccination, and at 124 days after the last vaccination. For Groups A, B, D, E: Day 1, Day 8, 29, 36, 57, 64, 85, and Day 181. For Group C: Day 1, Day 8, 29, 36, 57, 180, 187, 208, and Day 304.
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer of serum antibodies
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
titer of serum antibodies
  Day 1 (Pre-Dose 1) | 24.659 [9.006 to 67.515] | 29.209 [13.278 to 64.256] | 74.704 [19.641 to 284.138] | 29.884 [9.794 to 91.185] | 26.235 [15.640 to 44.008]
  Day 8 | 22.668 [11.176 to 45.978] | 26.915 [11.785 to 61.469] | 66.900 [16.501 to 271.230] | 28.233 [8.652 to 92.135] | 16.887 [7.941 to 35.908]
  Day 29: number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
  Day 29 | 32.515 [11.989 to 88.182] | 34.058 [11.830 to 98.049] | 139.103 [31.427 to 615.702] | 44.900 [10.445 to 193.011] | 49.354 [29.289 to 83.162]
  Day 36: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  Day 36 | 120.194 [37.282 to 387.497] | 226.177 [85.980 to 594.975] | 1079.771 [406.714 to 2866.647] | 489.783 [136.234 to 1760.843] | 420.482 [159.039 to 1111.705]
  Day 57: number analyzed (Participants) | 9 | 9 | 9 | 9 | 8
  Day 57 | 228.496 [91.931 to 567.934] | 868.743 [249.759 to 3021.767] | 2691.534 [1022.427 to 7085.447] | 868.512 [114.784 to 6571.573] | 1659.587 [538.253 to 5116.973]
  Day 64: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 64 | 498.632 [233.502 to 1064.803] | 1475.325 [528.085 to 4121.657] |  | 4062.047 [551.805 to 29902.258] | 3620.347 [1234.793 to 10614.663]
  Day 85: number analyzed (Participants) | 9 | 9 | 0 | 8 | 8
  Day 85 | 1186.982 [367.503 to 3833.783] | 4254.894 [1788.090 to 10124.837] |  | 4073.814 [589.783 to 28139.074] | 4479.711 [1703.143 to 11782.807]
  Day 180: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 180 |  |  | 376.322 [113.170 to 1251.378] |  |
  Day 181: number analyzed (Participants) | 9 | 9 | 0 | 6 | 8
  Day 181 | 514.170 [175.850 to 1503.385] | 1412.534 [626.880 to 3182.829] |  | 439.870 [105.239 to 1838.540] | 985.714 [364.226 to 2667.659]
  Day 187: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 187 |  |  | 2610.156 [844.732 to 8065.173] |  |
  Day 208: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 208 |  |  | 16343.056 [5920.195 to 45115.994] |  |
  Day 304: number analyzed (Participants) | 0 | 0 | 9 | 0 | 0
  Day 304 |  |  | 1471.551 [457.904 to 4729.075] |  |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs), MAAEs, NOCMCs, and PIMMCs were collected from the time of first study product injection through approximately 12 months after the last study product injection. Solicited AEs were collected from the time of each study product injection through 7 days after each study product injection. Unsolicited AEs were collected from the time of each study product injection through 28 days after the study product injection.
Arm/Group | Group A: 100 ug Sm-p80 Unadjuvanted | Group B: 10 ug Sm-p80 + GLA-SE | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster | Group D: 30 ug Sm-p80 + GLA-SE | Group E: 100 ug Sm-p80 + GLA-SE
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 100 ug Sm-p80 Unadjuvanted (N=9) | Group B: 10 ug Sm-p80 + GLA-SE (N=9) | Group C: 30 ug Sm-p80 + GLA-SE Delayed Booster (N=9) | Group D: 30 ug Sm-p80 + GLA-SE (N=9) | Group E: 100 ug Sm-p80 + GLA-SE (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (6) | 1 (2) | 4 (4) | 2 (4) | 3 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (6)
Fatigue (General disorders) | 8 (16) | 5 (6) | 7 (16) | 6 (7) | 5 (15)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 9 (26) | 8 (22) | 9 (22) | 8 (18) | 9 (20)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 3 (5) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Injection site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (4) | 3 (4) | 5 (6) | 3 (6) | 4 (6)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Platelet count increased (Investigations) | 0 (0) | 2 (6) | 2 (2) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1) | 6 (11) | 4 (6) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (12) | 6 (11) | 7 (17) | 5 (7) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT05292391/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05292391/SAP_001.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05292391/ICF_000.pdf